CLINICAL TRIAL: NCT03884465
Title: A Two Part, Phase 2 Open-label, Multi-Centre, Dose Escalation Hemodynamic Study to Evaluate Dose-Response and Safety of Inhaled LIQ861 (Treprostinil) in Pulmonary Arterial Hypertension (WHO Group 1) Subjects
Brief Title: Hemodynamic Evaluation of Dose-response and Safety of Dry Powder Inhalation of Treprostinil
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: COVID
Sponsor: Liquidia Technologies, Inc. (Industry)
Collaborators: FGK Clinical Research GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LTI-201; 2018-003414-40 (EudraCT Number)
Record Dates: First submitted 2019-03-04; First posted 2019-03-21 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary arterial hypertension; Pulmonary hypertension; PAH; PH; WHO Group 1 pulmonary arterial hypertension; WHO Group 1 pulmonary hypertension; WHO Group 1 PAH; WHO Group 1 PH; WHO Group 1; Group 1 PAH; Group 1 PH; Idiopathic PAH; Heritable PAH; Drug induced PAH; Toxin induced PAH; Pulmonary shunt; Idiopathic pulmonary arterial hypertension; Heritable pulmonary arterial hypertension; Drug induced pulmonary arterial hypertension; Toxin induced pulmonary arterial hypertension; Connective tissue disease
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary; Familial Primary Pulmonary Hypertension; Connective Tissue Diseases

STUDY DESIGN:
Intervention Model Description: Subjects will be enrolled in 4 sequential cohorts, each with an increasing initial dose of inhaled dry powder treprostinil (LIQ861) at 25μg, 50μg, 75μg, and 100μg capsule strengths (8 subjects at each dose level). Subjects will undergo right heart catheterization (RHC) at Day 1 to assess hemodynamic response.
  Subjects enrolled in Germany will continue in a follow-up hemodynamic and long-term safety study beginning immediately after the conclusion of the post-RHC assessments on Day 1 of Part A. Subjects will continue on therapy at four times daily (QID) on Day 1 and until Week 16 and may be titrated up or down by no more than one 25 μg increment per week, based upon symptomatic relief or side effects experienced by the subject. Investigators may also initiate Part B dosing at 25 μg before following this titration schedule.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Inhaled dry powder treprostinil (LIQ861) (Experimental): Full study population receives inhaled dry powder treprostinil (LIQ861) at 25μg, 50μg, 75μg or 100μg capsule strengths.
  Interventions: Drug: Inhaled dry powder treprostinil (LIQ861)

INTERVENTIONS:
Drug: Inhaled dry powder treprostinil (LIQ861) — Inhaled dry powder treprostinil (LIQ861) at 25μg, 50μg, 75μg, or 100μg capsule strengths. Single dose in the acute setting. QID in the chronic setting.
  Other Names: Inhaled treprostinil; Inhaled prostacyclin

SUMMARY:
Acute and chronic hemodynamic dose-response and safety evaluation of LIQ861 in PAH subjects.

DETAILED DESCRIPTION:
Data will be collected on acute and chronic hemodynamic response to inhaled dry powder treprostinil (LIQ861) via right-heart catheterization. Study subjects will contribute to the overall safety profile of LIQ861.

ELIGIBILITY:
Inclusion Criteria (A subject will be eligible for inclusion in this study only if all of the following criteria are met):

1. An Institutional Review Board (IRB) approved informed consent is signed and dated by the subject prior to any study related activities.
2. The subject is 18 years of age or older.
3. If the subject is a female of childbearing potential, then the subject has a negative pregnancy test at the Day 1 Visit (tests performed within 2 days before Day 1 are accepted) and agrees to practice a highly effective (failure rate of less than 1% per year when used consistently and correctly) method of birth control until 24 hours after completion of all study assessments defined in Appendix 1. If the subject is postmenopausal or has documented surgical sterilization, a pregnancy test and birth control is not necessary. It is the Investigator's responsibility for determining whether the subject has adequate birth control for study participation.
4. The subject has been diagnosed with PAH belonging to one of the following subgroups of the updated Nice Clinical Classification Group 1, which includes:

   1. Idiopathic PAH (1.1), or
   2. Heritable PAH (1.2), or
   3. Drug and toxin induced PAH (1.3), or
   4. PAH associated with connective tissue disease (1.4.1), HIV infection (1.4.2), or congenital heart disease (1.4.4) with simple systemic-to-pulmonary shunt at least 1 year after surgical repair
5. The subject is NYHA Functional Class II - IV at Screening and:

   1. has not previously been treated for PAH, or
   2. has documented stable doses of no more than 2 approved non prostacyclin PAH-disease specific therapies for at least 3 months prior to Screening, is willing and able to add LIQ861 to their treatment regimen and is willing to hold the dosing of these therapies for at least 12 hours prior to study-mandated right heart catheterization procedures.
6. The subject can complete a baseline six-minute walk distance (6MWD) ≥150 m.
7. The subject has had evidence of Forced Expiratory Volume in 1 Second (FEV1) and Forced Vital Capacity (FVC) ≥60% of predicted values and FEV1/FVC ratio ≥60% during the 6 month period prior to consent.

Exclusion Criteria (A subject is not eligible for inclusion in the study if any of the following criteria apply):

1. The subject's clinical condition is such that, in the opinion of the Investigator, they are not expected to remain clinically stable for the duration of the study.
2. Subjects with pulmonary hypertension (PH) in the Updated Nice Classification Groups 2-5, or PAH Group 1 subgroups not covered by the inclusion criteria (e.g., associated with portal hypertension [1.4.3] or with schistosomiasis [1.4.5]).
3. The subject is currently taking prostacyclin analogues or agonists, including treprostinil, iloprost, epoprostenol or selexipag.
4. The subject has discontinued any medication (except for anticoagulants, but otherwise including but not limited to oxygen, a different class of vasodilator, diuretic, digoxin, and digitalis) for pulmonary hypertension within 14 days prior to Day 1.
5. The subject has had a new type of therapy (including but not limited to oxygen, a different class of vasodilator, diuretic, digoxin, and digitalis) for pulmonary hypertension added within 30 days prior to Day 1.
6. The subject has uncontrolled systemic hypertension as evidenced by systolic blood pressure greater than 160 mmHg or diastolic blood pressure greater than 100 mmHg at the time of screening.
7. The subject has a history of hemodynamically significant left-sided heart disease including, but not limited to: aortic or mitral valve disease, pericardial constriction, restrictive or congestive cardiomyopathy, or symptomatic coronary artery disease (CAD).
8. The subject has had an atrial septostomy.
9. The subject has a history of prolongation of QT interval on ECG as follows: Male subjects with a corrected QT interval using Fridericia's formula (QTcF) >450 msec and female subjects with QTcF >470 msec.
10. The subject has any serious or life-threatening disease other than conditions associated with PAH.
11. The subject is taking any excluded medications listed in the Investigator's Brochure, namely inhibitors and inducers of CYP2C8 (see Appendix 3).
12. The subject has a hypersensitivity or allergy to any of the ingredients of LIQ861, NO, or other clinically relevant allergies (clinical relevance per Investigator judgment).
13. The subject has had an acute pulmonary embolus within 6 months prior to Baseline.
14. The subject has had a stroke or transient ischemic attack within 6 months prior to Baseline.
15. The subject has evidence of an active uncontrolled sepsis or systemic infection in the period after informed consent up to Baseline.
16. The subject is pregnant or lactating.
17. The subject has any musculoskeletal disease or any other disease that limits evaluation of 6MWD.
18. The subject has participated in an investigational product or device study within the 30 days prior to Baseline.
19. The subject has current evidence of drug abuse in the opinion of the Investigator.
20. The subject has severe hepatic impairment as evidenced by any history of ascites AND encephalopathy.
21. The subject has severe renal impairment (estimated glomerular filtration rate [eGFR] <35 mL/min utilizing the Modification of Diet in Renal Disease (MDRD) study equation or requires dialytic support.
22. The subject is an employee or an immediate family member to an employee of the Sponsor or the Investigator.
23. The subject is not a member or beneficiary of a social security scheme.
24. The subject lacks a legal protection measure.
25. The subject has been deprived of their liberty by a judicial or administrative decision.
26. The subject has a known Hepatitis B or Hepatitis C infection with active viral replication.
27. The subject has a known HIV infection with CD4 count less than 200 and more than undetectable viral load, defined as less than 50 copies /mL.
28. The subject required use of intravenous inotropes including, but not limited to, Levosimendan, Dopamine, Dobutamine, Dopexamine, Epinephrine, Isoprenaline (isoproterenol), Norepinephrine (noradrenaline), Milrinone, or Amrinone, within 30 days prior to Baseline.
29. The subject required intravenous diuretic therapy within 30 days prior to Baseline.
30. Subjects taking vitamin K antagonist therapy with a known INR ≥3.5 (assessed per local care standards) at the time of screening assessments or at Baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2020-12-23 (Actual); Study Completion 2020-12-23 (Actual)

PRIMARY OUTCOMES:
Change in Pulmonary Vascular Resistance (PVR) | 2 hours (120 minutes) post-dose on Day 1 and Week 16
  Calculated in Wood units
Change in Pulmonary Artery Pressure (PAP) | 2 hours (120 minutes) post-dose on Day 1 and Week 16
  Systolic, diastolic, and mean pressure measured in millimeters of mercury (mmHG)
Change in Cardiac Output (CO) | 2 hours (120 minutes) post-dose on Day 1 and Week 16
  Measured in liters per minute (L/min)
Change in Pulmonary Artery Oxygen Saturation (PAO2%) | 2 hours (120 minutes) post-dose on Day 1 and Week 16
  Measured as a percent oxyhemoglobin saturation

SECONDARY OUTCOMES:
Number of participants with treatment emergent adverse events (AEs) | Baseline until the end of study, approximately 18 months (Mar-2021)
  Treatment-emergent adverse events and serious adverse events will be grouped by MedDRA System Organ Class, dose level at onset, time on drug at onset, and relationship to dose titration.

CONTACTS AND LOCATIONS:
Overall Officials: Ardeschir Ghofrani, Prof. MD., Principal Investigator — Universitatskinikum Giessen und Marburg GmbH
Locations (3):
- France (2):
  - CHRU de Nancy, Nancy, Vandoeuvre Les Nancy
  - CHU de Bicetre, Le Kremlin-Bicêtre
- Studienambulanz fur Pulmonale Hypertonie at Medizinishe Klinik II, Universitatskinikum Giessen und Marburg GmbH, Giessen, Germany

IPD SHARING:
Plan to Share IPD: Undecided